CLINICAL TRIAL: NCT07093008
Title: A Phase 1, Investigator- and Participant-blinded, Placebo-Controlled, Randomized, Crossover Study to Assess the Relative Bioavailability of Two Formulations of AQ280 in Healthy Participants
Brief Title: Comparing the Extent to Which AQ280 is Made Available in the Body After Single Oral Doses of a Capsule Formulation Versus a Tablet for Oral Suspension Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AQILION AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ARIA-2
Record Dates: First submitted 2025-07-04; First posted 2025-07-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Suspensions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intervention Sequence 1 (Placebo Comparator): Treatment Period 1: Placebo Capsule will be administered orally.
  Treatment Period 2: Placebo Tablet for Oral Suspension will be administered orally.
  Interventions: Drug: Placebo Capsule; Drug: Placebo Tablet for Oral Suspension
- Intervention Sequence 2 (Placebo Comparator): Treatment Period 1: Placebo Tablet for Oral Suspension will be administered orally.
  Treatment Period 2: Placebo Capsule will be administered orally.
  Interventions: Drug: Placebo Capsule; Drug: Placebo Tablet for Oral Suspension
- Intervention Sequence 3 (Experimental): Treatment Period 1: AQ280 Capsule will be administered orally.
  Treatment Period 2: AQ280 Tablet for Oral Suspension will be administered orally.
  Interventions: Drug: AQ280 Capsule; Drug: AQ280 Tablet for Oral Suspension
- Intervention Sequence 4 (Experimental): Treatment Period 1: AQ280 Tablet for Oral Suspension will be administered orally.
  Treatment Period 2: AQ280 Capsule will be administered orally.
  Interventions: Drug: AQ280 Capsule; Drug: AQ280 Tablet for Oral Suspension

INTERVENTIONS:
Drug: AQ280 Capsule — AQ280 administered orally in capsule formulation.
  Arms: Intervention Sequence 3; Intervention Sequence 4
Drug: AQ280 Tablet for Oral Suspension — AQ280 administered orally in tablet for oral suspension formulation.
  Arms: Intervention Sequence 3; Intervention Sequence 4
Drug: Placebo Capsule — Placebo administered orally in capsule formulation.
  Arms: Intervention Sequence 1; Intervention Sequence 2
Drug: Placebo Tablet for Oral Suspension — Placebo administered orally in tablet for oral suspension formulation.
  Arms: Intervention Sequence 1; Intervention Sequence 2

SUMMARY:
This is a Phase 1, investigator- and participant-blinded, placebo-controlled, randomized, crossover study to compare bioavailability of AQ280 following single oral doses of a capsule formulation versus a tablet for oral suspension formulation in healthy participants.

ELIGIBILITY:
Inclusion Criteria -

1. Male or female, of any race, between 18 and 65 years of age, inclusive.

   1. Females must not be pregnant or lactating.
   2. Males and females of childbearing potential must agree to use contraception
2. Body mass index between 18.0 and 29.9 kg/m2, inclusive.
3. In good health, as determined by no clinically significant findings from medical history, 12-lead ECG and vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in, and from the physical examination at check-in, as assessed by the investigator or designee.
4. Able to comprehend and are willing to sign the ICF and abide by the study restrictions.

Exclusion Criteria -

An individual who meets any of the following criteria at screening, unless otherwise stated, will be excluded from participation in this study:

Medical Conditions

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator or designee.
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed).
4. Any of the following:

   1. QTcF >450 ms in males or >470 ms in females, based on the longest value from the triplicate ECG measurements
   2. QRS duration >120 ms, based on the longest value from the triplicate ECG measurements
   3. PR interval >210 ms, based on the longest value from the triplicate ECG measurements
   4. findings which would make QTc measurements difficult or QTc data uninterpretable
   5. history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia, or family history of long QT syndrome).
5. Participants with an increased risk of thromboembolic events (eg, history of recurrent venous thrombosis or Factor V Leiden mutation).
6. Magnesium < LLN; participants with values that are borderline < LLN may be included, as determined by the investigator or designee.
7. History of any significant infectious disease, as assessed by the investigator, within 2 weeks prior to the first dose of IMP.
8. AST and/or ALT values > 1.2 × ULN.
9. Congenital nonhemolytic hyperbilirubinemia.
10. Hemoglobin value, neutrophil count (absolute), lymphocyte count (absolute), and/or platelet count < LLN; participants with values that are borderline < LLN may be included, as determined by the investigator or designee.
11. White blood cell count > ULN; participants with values that are borderline > ULN may be included, as determined by the investigator or designee.
12. eGFR < 90 mL/min/1.73 m2 (calculated using the CKD-EPI equation3).
13. Significant history of herpes infection (ie, severe herpes outbreaks requiring anti-viral treatment).
14. Positive hepatitis panel and/or positive human immunodeficiency virus test. Participants whose results are compatible with prior immunization may be included.
15. Current active tuberculosis based on Quantiferon™ tuberculosis Gold test or history of latent infection.

    Prior and Concomitant Therapy
16. Administration of any vaccine within 30 days prior to dosing.
17. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
18. Use or intend to use any prescription medications/products, other than hormone replacement therapy, oral, implantable, transdermal, injectable, intravaginal, or intrauterine contraceptives, within 14 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
19. Use or intend to use any slow-release medications/products considered to still be active within 14 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
20. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.

    Prior and Concurrent Clinical Study Experience
21. Participation in a clinical study involving administration of an IMP (new chemical entity) in the past 90 days or 5 half-lives of that drug (if known) prior to dosing, whichever is longer.
22. Have previously completed or withdrawn from this study or any other study investigating AQ280 and have previously received AQ280.

    Diet and Lifestyle
23. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
24. Positive urine drug screen at screening. Positive alcohol test result or positive urine drug screen at check-in.
25. History of alcoholism or drug/chemical abuse within 2 years prior to check-in.

    Other
26. Use of tobacco- or nicotine-containing products within 3 months prior to check-in.
27. Receipt of blood products within 2 months prior to check-in.
28. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
29. Poor peripheral venous access.
30. Participants who, in the opinion of the investigator or designee, should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability (Frel) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Maximum observed concentration (Cmax) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Time of the maximum observed concentration (Tmax) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Apparent terminal elimination half-life (t1/2) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Apparent total clearance (CL/F) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Apparent volume of distribution during the terminal phase (Vz/F) | Pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)

SECONDARY OUTCOMES:
Incidence and severity of adverse events | From screening up to end of study (approximately 7 weeks)
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Screening, Day -1 and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Number of participants with abnormal electrocardiograms | Screening, Day -1, pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
  QTcF interval of >500 msec or change from baseline (Day 1, predose) >60 msec
Number of participants with clinically significant abnormalities in vital signs - blood pressure (systolic in mm Hg) | Screening, Day -1, pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Number of participants with clinically significant abnormalities in vital signs - blood pressure (diastolic in mm Hg) | Screening, Day -1, pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Number of participants with clinically significant abnormalities in vital signs - pulse rate (beats per minute) | Screening, Day -1, pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Number of participants with clinically significant abnormalities in vital signs - oral body temperature (°C) | Screening, Day -1, pre dose and up to 48 hours post dose (up to end of study - approximately 7 weeks)
Incidence of abnormal physical examinations | From screening up to end of study (approximately 7 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Törnell, Study Director — AQILION AB
Locations (1):
- Clinical Research Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No